CLINICAL TRIAL: NCT00680901
Title: A Phase III Study for ErbB2 Positive Advanced or Metastatic Gastric, Esophageal, or Gastroesophageal Junction Adenocarcinoma Treated With Capecitabine Plus Oxaliplatin With or Without Lapatinib
Brief Title: LOGiC - Lapatinib Optimization Study in ErbB2 (HER2) Positive Gastric Cancer: A Phase III Global, Blinded Study Designed to Evaluate Clinical Endpoints and Safety of Chemotherapy Plus Lapatinib
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGF110656; 2007-005725-29 (EudraCT Number); CLAP016C2301 (Other: Novartis)
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Results first posted 2013-10-29 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Neoplasms, Gastrointestinal Tract
Keywords: unresectable; HER2; ErbB2; TYKERB; capecitabine; CapeOx; gastric/esophageal cancer; GE junction; metastatic; lapatinib; oxaliplatin
MeSH Terms: conditions — Neoplasms; Esophageal Neoplasms; Neoplasm Metastasis | interventions — Lapatinib; Capecitabine; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CapeOx plus Lapatinib (Experimental): CapeOx plus Lapatinib
  Interventions: Drug: Lapatinib; Drug: Capecitabine; Drug: Oxaliplatin
- CapeOx plus Placebo (Placebo Comparator): CapeOx plus Placebo
  Interventions: Drug: Placebo; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Lapatinib — 5 pills at 250mg each once daily
  Other Names: Tykerb
  Arms: CapeOx plus Lapatinib
Drug: Placebo — 5 pills once daily
  Arms: CapeOx plus Placebo
Drug: Capecitabine — 1700mg/m2/day in two daily doses
Drug: Oxaliplatin — 130mg/m2 on day 1

SUMMARY:
This was an international multi-center trial that enrolled patients with locally advanced, unresectable, or metastatic gastric, esophageal, or gastro-esophageal junction cancer whose tumors had amplification of the ErbB2 (HER2) gene. The trial investigated whether lapatinib, when added to the chemotherapy regimen, capecitabine plus oxaliplatin (CapeOx), extended the time to progression and overall survival. Tumor ErbB2 (HER2) status had to be known before trial entry. CapeOx was administered to all patients, and patients were randomly assigned to receive either lapatinib or placebo.

ELIGIBILITY:
Key inclusion criteria:

* Histologically confirmed gastric adenocarcinoma or adenocarcinoma of the esophagus or gastro-esophageal junction.
* Gastric cancer that is unresectable due to locally advanced (defined as stage IV: T4N1-3 or TanyN3), metastatic, or locally recurrent disease; Esophageal cancer that is unresectable due to locally advanced (T3N1 or T4Nany), metastatic or locally recurrent disease.
* Measurable or non-measurable, but radiologically evaluable disease, according to RECIST.
* HER2 amplification by FISH assessed by the local or designated central laboratory; Subjects with unknown HER2 status were not eligible.
* Adequate organ function, as defined in the study protocol, assessed within 14 days prior randomization.
* Cardiac ejection fraction within institutional range of normal as measured by echocardiogram (ECHO).
* Prior/Concurrent Therapy:

  * At least 3 weeks following major surgery, such as gastrectomy, and were recovered from any related toxicity More than 5 years since prior chemotherapy for malignancy other than GC. At least 4 weeks since prior radiotherapy
  * More than 5 years since prior biologic or hormonal therapy or immunotherapy for malignancy other than gastric carcinoma.

Key exclusion criteria:

* Pregnant or lactating females at any time during the study.
* Known history of active CNS disease.
* Uncontrolled ascites.
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy other than for pain relief, immunotherapy, biologic therapy, hormonal therapy or surgery) while taking investigational treatment.
* Gastric carcinoid, epidermoid, sarcomas, or squamous cell carcinoma.
* Prior palliative chemotherapy for the treatment of gastric cancer.
* Prior treatment with oxaliplatin-based neoadjuvant or adjuvant chemotherapy completed <12 months.
* Malabsorption syndrome or uncontrolled inflammatory gastrointestinal disease (such as Crohn's disease or ulcerative colitis).
* Known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure.
* Uncontrolled infection.
* History of other malignancy. However, subjects who were disease-free for 5 years, or subjects with a history of a completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, were eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2008-06-04 (Actual); Primary Completion 2012-09-24 (Actual); Study Completion 2024-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (158):
- United States (10):
  - Novartis Investigative Site, Alhambra, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, La Verne, California
  - Novartis Investigative Site, Northridge, California
  - Novartis Investigative Site, Oxnard, California
  - Novartis Investigative Site, Redondo Beach, California
  - Novartis Investigative Site, Santa Maria, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Terre Haute, Indiana
  - Novartis Investigative Site, Henderson, Nevada
- Argentina (9):
  - Novartis Investigative Site, Ciudad Aut6noma de Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, Neuquén, Neuquén Province
  - Novartis Investigative Site, Cipolletti, Río Negro Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, La Rioja
  - Novartis Investigative Site, San Miguel de Tucumán
  - Novartis Investigative Site, Santa Fe
- Brazil (8):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Florianópolis, Santa Catarina
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, Jaú, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Rio de Janeiro
- Canada (6):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Saint John, New Brunswick
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Chile (4):
  - Novartis Investigative Site, Temuco, Región de La Araucania
  - Novartis Investigative Site, Viña del Mar, Región de Valparaíso
  - Novartis Investigative Site, Santiago, Región Metro de Santiago
  - Novartis Investigative Site, Santiago
- China (12):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Fuzhou
  - Novartis Investigative Site, Hangzhou
  - Novartis Investigative Site, Qingdao
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Hong Kong (2):
  - Novartis Investigative Site, Pokfulam
  - Novartis Investigative Site, Tuenmen
- Hungary (7):
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Kecskemét
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szolnok
- India (8):
  - Novartis Investigative Site, Coimbatore
  - Novartis Investigative Site, Kochi
  - Novartis Investigative Site, Kolkata
  - Novartis Investigative Site, Nagpur
  - Novartis Investigative Site, New Delhi
  - Novartis Investigative Site, Pārel
  - Novartis Investigative Site, Pune
  - Novartis Investigative Site, Trivandrum
- Israel (8):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Zrifin
- Italy (17):
  - Novartis Investigative Site, L’Aquila, Abruzzo
  - Novartis Investigative Site, Bari, Apulia
  - Novartis Investigative Site, Rionero in Vulture (PZ), Basilicate
  - Novartis Investigative Site, Cesena, Emilia-Romagna
  - Novartis Investigative Site, Meldola (FC), Emilia-Romagna
  - Novartis Investigative Site, Modena, Emilia-Romagna
  - Novartis Investigative Site, Parma, Emilia-Romagna
  - Novartis Investigative Site, Piacenza, Emilia-Romagna
  - Novartis Investigative Site, Rimini, Emilia-Romagna
  - Novartis Investigative Site, Udine, Friuli Venezia Giulia
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Genoa, Liguria
  - Novartis Investigative Site, Bergamo, Lombardy
  - Novartis Investigative Site, Treviglio (BG), Lombardy
  - Novartis Investigative Site, Pesasro, The Marches
  - Novartis Investigative Site, Florence, Tuscany
  - Novartis Investigative Site, Macerata
- Mexico (3):
  - Novartis Investigative Site, Acapulco de Juárez, Guerrero
  - Novartis Investigative Site, Mexico City
  - Novartis Investigative Site, Oaxaca City
- Netherlands (3):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Nijmegen
- Peru (2):
  - Novartis Investigative Site, Callao
  - Novartis Investigative Site, Lima
- Poland (10):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Płock
  - Novartis Investigative Site, Rybnik
  - Novartis Investigative Site, Szczecin
  - Novartis Investigative Site, Słupsk
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, San Juan, Puerto Rico
- Russia (11):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Kursk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Sochi
  - Novartis Investigative Site, Stavropol
  - Novartis Investigative Site, Ufa
- South Korea (7):
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Hwasun
  - Novartis Investigative Site, Seodaemun-gu, Seoul
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Suwon
  - Novartis Investigative Site, Suwon, Kyonggi-do
- Taiwan (3):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Hatyai, Songkhla
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Gaziantep
  - Novartis Investigative Site, Trabzon
- Ukraine (20):
  - Novartis Investigative Site, Cherkasy
  - Novartis Investigative Site, Chernivtsi
  - Novartis Investigative Site, Dnipro
  - Novartis Investigative Site, Dnipropetrovsk
  - Novartis Investigative Site, Donetsk
  - Novartis Investigative Site, Ivano-Frankivsk
  - Novartis Investigative Site, Kharkiv
  - Novartis Investigative Site, Kryvyi Rih
  - Novartis Investigative Site, Kyiv
  - Novartis Investigative Site, Lutsk
  - Novartis Investigative Site, Lviv
  - Novartis Investigative Site, Odesa
  - Novartis Investigative Site, Plyuty
  - Novartis Investigative Site, Simferopil
  - Novartis Investigative Site, Simferopol
  - Novartis Investigative Site, Sumy
  - Novartis Investigative Site, Ternopil
  - Novartis Investigative Site, Uzhhorod
  - Novartis Investigative Site, Vinnitsia
  - Novartis Investigative Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Chu MP, Hecht JR, Slamon D, Wainberg ZA, Bang YJ, Hoff PM, Sobrero A, Qin S, Afenjar K, Houe V, King K, Koski S, Mulder K, Hiller JP, Scarfe A, Spratlin J, Huang YJ, Khan-Wasti S, Chua N, Sawyer MB. Association of Proton Pump Inhibitors and Capecitabine Efficacy in Advanced Gastroesophageal Cancer: Secondary Analysis of the TRIO-013/LOGiC Randomized Clinical Trial. JAMA Oncol. 2017 Jun 1;3(6):767-773. doi: 10.1001/jamaoncol.2016.3358. PMID 27737436
- [Derived] Hecht JR, Bang YJ, Qin SK, Chung HC, Xu JM, Park JO, Jeziorski K, Shparyk Y, Hoff PM, Sobrero A, Salman P, Li J, Protsenko SA, Wainberg ZA, Buyse M, Afenjar K, Houe V, Garcia A, Kaneko T, Huang Y, Khan-Wasti S, Santillana S, Press MF, Slamon D. Lapatinib in Combination With Capecitabine Plus Oxaliplatin in Human Epidermal Growth Factor Receptor 2-Positive Advanced or Metastatic Gastric, Esophageal, or Gastroesophageal Adenocarcinoma: TRIO-013/LOGiC--A Randomized Phase III Trial. J Clin Oncol. 2016 Feb 10;34(5):443-51. doi: 10.1200/JCO.2015.62.6598. Epub 2015 Nov 30. PMID 26628478

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 186 centers in 21 countries in North America (Canada and US), Asia (China, Hong Kong, Korea and Taiwan), and Rest of World (ROW) (Argentina, Brazil, Chile, Estonia, Hungary, India, Israel, Italy, Mexico, Netherlands, Peru, Poland, Russian Federation, Turkey, and Ukraine).
Pre-assignment Details: Participants were randomized into one of two treatment arms: CapeOx plus lapatinib (the experimental arm) or CapeOx plus placebo (the control arm) using a 1:1 randomization.
Groups:
- CapeOx Plus Lapatinib: Participants received a combination therapy consisting of:
  1. Oxaliplatin (Ox): 130 mg/m² intravenously on Day 1 of each 21-day cycle, for up to 8 cycles.
  2. Capecitabine (Cape): 1700 mg/m² per day, taken orally in two divided doses from the evening of Day 1 to the morning of Day 15 (28 doses per cycle), followed by a minimum 6.5-day rest period. The dose could be increased to 2000 mg/m²/day after the first cycle at the investigator's discretion.
  3. Lapatinib: 1250 mg orally once daily, starting on Day 1 and continued daily throughout the cycle, including the rest period.
  After discontinuing oxaliplatin, capecitabine and lapatinib were continued until disease progression, unacceptable toxicity, or withdrawal of consent.
- CapeOx Plus Placebo: Participants received a combination therapy consisting of:
  1. Oxaliplatin (Ox): 130 mg/m² intravenously on Day 1 of each 21-day cycle, for up to 8 cycles.
  2. Capecitabine (Cape): 1700 mg/m² per day, taken orally in two divided doses from the evening of Day 1 to the morning of Day 15 (28 doses per cycle), followed by a minimum 6.5-day rest period. The dose could be increased to 2000 mg/m²/day after the first cycle at the investigator's discretion.
  3. Lapatinib matching placebo: Taken orally once daily starting on Day 1 and continued throughout each cycle, including the rest period.
  After discontinuing oxaliplatin, capecitabine and the lapatinib placebo were continued until disease progression, unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Started (The Intent-to-Treat (ITT) population included all subjects who had been randomized to study treatment, regardless of whether they actually received the study medication.) | 272 | 273
Primary Efficacy (PE) Population (The Primary Efficacy (PE) population included all randomized subjects with centrally confirmed HER2-positive tumors based on FISH assessment. This population was used to analyze efficacy and health outcomes at the time of the primary CSR.) | 249 | 238
Safety Population (The Safety population included all randomized subjects who had received at least one dose of study medication. Analyses were based on the actual treatment received, and this population was used for the final safety analysis.) | 270 | 267
Ongoing: On Study Treatment (Due to local regulations in China (HGRAC), data collection at all sites in China was immediately stopped as of 01-Jul-2016. No data from Chinese subjects was transferred or processed thereafter. Consequently, this subject was marked as "ongoing" in the database.) | 1 | 0
Ongoing: In Follow Up (Due to local regulations in China, data from Chinese subjects dated from 01-Jul-2016 onward was excluded. As noted in the primary CSR, the subject had been withdrawn from the study on 05 Apr 2011 due to being lost to follow-up, and overall survival was unknown. However, a data transition issue from the previous database (TRIO) led to the subject being incorrectly reported as "ongoing".) | 1 | 0
Completed | 243 | 233
Not Completed | 29 | 40
Not completed — Ongoing: On Study Treatment | 1 | 0
Not completed — Ongoing: In Follow Up | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 3 | 5
Not completed — Subject decided to withdraw from the study | 4 | 15
Not completed — Sponsor decision | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Subject reached protocol defined stopping criteria | 1 | 0
Not completed — Other protocol defined stopping criteria | 17 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo | Total
Number analyzed (Participants) | 272 | 273 | 545
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (11.20) | 58.5 (11.23) | 58.9 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 73 | 139
  Male | 206 | 200 | 406
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage (Hrtg) | 2 | 3 | 5
  American Indian or Alaska Native | 3 | 3 | 6
  Central/South Asian Hrtg | 11 | 3 | 14
  Japanese/East Asian Hrtg/South East Asian Hrtg | 112 | 114 | 226
  White | 144 | 150 | 294

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at the Time of Primary Analysis
Description: Overall Survival was defined as the time from randomization to death from any cause. Participants who had not died were censored at their follow-up visit, either because follow-up had ended or was still ongoing.
Time Frame: From date of randomization till death due to any cause, assessed up the cut-off date for Primary Analysis (24-Sep-2012) (average of 4 years)
Population: Primary Efficacy (PE) population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 249 | 238
Months | 12.2 [10.6 to 14.2] | 10.5 [9.0 to 11.3]
Statistical Analysis 1: Comparison: CapeOx Plus Lapatinib vs CapeOx Plus Placebo; Primary Analysis: OS (PE population); Test type: Superiority or Other; p = 0.3492, Log Rank — Stratified log-rank test was conducted stratifying for prior adjuvant/neo-adjuvant treatment use and region; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.73 to 1.12] — Pike estimator of HR was based on the stratified log rank test

2. Primary Outcome: Overall Survival in All Randomized Participants at the Time of Primary Analysis
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Intent-to-Treat (ITT) Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 272 | 273
Months | 11.9 [10.4 to 13.8] | 10.4 [9.1 to 11.3]
Statistical Analysis 1: Comparison: CapeOx Plus Lapatinib vs CapeOx Plus Placebo; Primary Analysis: OS (ITT population); Test type: Superiority or Other; p = 0.3244, Log Rank — Stratified log-rank test was conducted stratifying for prior adjuvant/neo-adjuvant treatment use and region; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.74 to 1.10] — Pike estimator of HR was based on the stratified log rank test

3. Secondary Outcome: Overall Survival at the Time of Final Analysis
Description: as for outcome 1
Time Frame: From date of randomization till death due to any cause, assessed up the cut-off date for Final Analysis (03-Oct-2024) (average of 16 years)
Population: Primary Efficacy (PE) population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 249 | 238
Months | 12.0 [10.4 to 13.8] | 10.4 [9.0 to 11.3]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-Free Survival (PFS) was defined as the time from randomization to the earliest occurrence of disease progression or death from any cause. Per RECIST v1.0, progression was defined as at least a 20% increase in the sum of diameters of target lesions from the smallest recorded sum or the appearance of one or more new lesions. Participants with symptomatic progression, even without radiological confirmation, were also counted. Those who had neither progressed nor died were censored at their follow-up visit, either because follow-up had ended or was ongoing. Participants who received non-study anti-cancer therapies before progression were also censored.
Time Frame: From date of randomization till the earliest date of disease progression or death due to any cause, assessed up the cut-off date for Final Analysis (03-Oct-2024) (average of 16 years)
Population: Primary Efficacy (PE) population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 249 | 238
Months | 6.2 [5.6 to 7.0] | 5.4 [4.4 to 5.7]

5. Secondary Outcome: Percentage of Participants With a Confirmed Complete Response (CR) or a Partial Response (PR)
Description: A participant was considered a responder if they had achieved either a complete response (CR), defined as the disappearance of all target and non-target lesions, or a partial response (PR), defined as at least a 30% reduction in the sum of the longest diameters of target lesions from baseline, as assessed by the investigator and confirmed by radiographic imaging within four weeks of the initial observation.
Time Frame: From date of randomization till the date of the first documented response of CR or PR, assessed up the cut-off date for Final Analysis (03-Oct-2024) (average of 16 years)
Population: Primary Efficacy (PE) population
Measure: Count of Participants; unit: Participants
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 249 | 238
Participants | 131 | 94

6. Secondary Outcome: Percentage of Participants With Clinical Benefit (CB)
Description: Clinical Benefit (CB) was defined as evidence of a complete response (CR), partial response (PR), or stable disease (SD). CR referred to the disappearance of all target and non-target lesions, PR to at least a 30% reduction in the sum of the longest diameters of target lesions from baseline, and SD to neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progression, based on the smallest sum of diameters recorded since treatment initiation. All assessments were made by the investigator.
Time Frame: From date of randomization till date of disease progression (PD) or death due to any cause, assessed up the cut-off date for Final Analysis (03-Oct-2024) (average of 16 years)
Population: Primary Efficacy (PE) population
Measure: Count of Participants; unit: Participants
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 249 | 238
Participants | 199 | 188

7. Secondary Outcome: Time to Response (TTR)
Description: Time to Response (TTR) was defined as the duration from randomization to the first documented evidence of either a complete response (CR) (the disappearance of all target and non-target lesions) or a partial response (PR) (at least a 30% reduction in the sum of the longest diameters of target lesions from baseline) as assessed by the investigator.
Time Frame: From date of randomization till the first documented evidence of confirmed CR or PR, assessed up the cut-off date for Final Analysis (03-Oct-2024) (average of 16 years)
Population: Primary Efficacy (PE) population. Only those participants who had a confirmed CR or PR were analyzed for time to response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 131 | 94
Months | 1.4 [1.4 to 1.5] | 1.4 [1.4 to 1.6]

8. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response (DOR) was defined as the time from the first documented evidence of a complete response (CR) or partial response (PR) until the first recorded sign of disease progression or death from any cause. According to RECIST, progression was defined as at least a 20% increase in the sum of diameters of target lesions from the smallest recorded sum or the appearance of one or more new lesions. Participants who had neither progressed nor died were censored at their follow-up visit, either because follow-up had ended or was ongoing. Those who received non-study anti-cancer therapies before progression were also censored.
Time Frame: From the time of the first documented evidence of a confirmed CR or PR until the earliest date of disease progression or death due to any cause, assessed up the cut-off date for Final Analysis (03-Oct-2024) (average of 16 years)
Population: Primary Efficacy (PE) population. Only those participants who had a confirmed CR or PR were analyzed for duration of response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 131 | 94
Months | 7.3 [6.4 to 8.5] | 5.6 [4.6 to 6.0]

9. Secondary Outcome: Percentage of Participants With Any On-therapy Adverse Event (AE) and Serious Adverse Event (SAE)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a participant that was temporally associated with the use of a medicinal product, regardless of its causal relationship. This included any unfavorable or unintended sign (such as abnormal lab findings), symptom, or disease, whether new or worsened. A Serious Adverse Event (SAE) was defined as any such occurrence that, at any dose, resulted in death, was life-threatening, required hospitalization or its prolongation, caused disability or incapacity, led to a congenital anomaly or birth defect, or was a potential case of drug-induced liver injury.
Time Frame: From the first dose of study medication until 30 days after the last dose, assessed up the cut-off date for Final Analysis (03-Oct-2024) (average of 16 years)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 270 | 267
Participants
  On-Therapy Adverse Events (Any AE regardless of seriousness) | 255 | 237
  On-Therapy Serious Adverse Events | 73 | 54

10. Secondary Outcome: Percentage of Participants With On-therapy Adverse Event (AE) by Maximum Grade
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a participant that was temporally associated with the use of a medicinal product, regardless of its relationship to the product. This included any unfavorable or unintended sign (such as abnormal lab results), symptom, or disease, whether new or worsened. The severity of AEs was graded according to NCI CTCAE version 3.0: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life-threatening), and Grade 5 (death related to toxicity).
Time Frame: as for outcome 9
Population: Safety population. Only participants with On-therapy AEs
Measure: Count of Participants; unit: Participants
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 255 | 237
Participants
  Grade 1 | 43 | 56
  Grade 2 | 85 | 78
  Grade 3 | 94 | 69
  Grade 4 | 17 | 25
  Grade 5 | 16 | 9

11. Secondary Outcome: Percentage of Participants With On-therapy Serious Adverse Event (SAE) by Maximum Grade
Description: A Serious Adverse Event (SAE) was defined as any such occurrence that resulted in death, was life-threatening, required hospitalization or its prolongation, caused disability or incapacity, led to a congenital anomaly or birth defect, or was a potential case of drug-induced liver injury. The severity of SAEs was graded according to NCI CTCAE version 3.0: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life-threatening), and Grade 5 (death related to toxicity).
Time Frame: as for outcome 9
Population: Safety population. Only participants with on-therapy Serious Adverse Events (SAEs)
Measure: Count of Participants; unit: Participants
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 73 | 54
Participants
  Grade 1 | 3 | 3
  Grade 2 | 6 | 4
  Grade 3 | 37 | 21
  Grade 4 | 13 | 18
  Grade 5 | 14 | 8

12. Secondary Outcome: Mean Change From Baseline in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life (QOL) Questionnaire Core 30 (QLQ-C30) Domain Scores
Description: The EORTC QLQ-C30 is a comprehensive questionnaire developed for assessing the quality of life of cancer patients across different aspects including function scales namely physical, role, cognitive, emotional and social; symptom scales such as fatigue, pain, nausea and vomiting; and a global scale pronouncing overall health status. Its scoring method involves a 4-point Likert scale (ranging from 1 'Not at all' to 4 'Very Much'). Domain scores are calculated by averaging the items within the respective domain and then linearly transforming the score to fit within a 0-100 scale to finalize the scores. In terms of interpretation, a high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Time Frame: From Baseline up to disease progression (PD), assessed up the cut-off date for Final Analysis (03-Oct-2024) (average of 16 years)
Population: Primary Efficacy (PE) population. Only those participants contributing data at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 61 | 61
Scores on a scale
  Global health status/QoL: number analyzed (Participants) | 61 | 60
  Global health status/QoL | -6.6 (24.63) | -5.1 (23.97)
  Physical functioning: number analyzed (Participants) | 60 | 61
  Physical functioning | -9.4 (25.61) | -9.6 (22.33)
  Role functioning: number analyzed (Participants) | 60 | 61
  Role functioning | -8.9 (34.64) | -11.7 (31.67)
  Emotional functioning | -3.8 (27.37) | -7.1 (23.61)
  Cognitive functioning | -7.4 (21.41) | -10.4 (21.98)
  Social functioning | -4.9 (32.54) | -0.5 (26.52)
  Fatigue | 5.5 (26.42) | 5.6 (25.30)
  Nausea and vomiting | 3.3 (27.69) | 4.4 (20.62)
  Pain | 4.9 (30.48) | 7.7 (30.06)
  Dyspnoea: number analyzed (Participants) | 60 | 60
  Dyspnoea | 6.7 (26.61) | 7.8 (27.70)
  Insomnia: number analyzed (Participants) | 61 | 60
  Insomnia | 0.0 (33.33) | 3.3 (35.09)
  Appetite loss | -0.5 (39.20) | 5.5 (37.11)
  Constipation: number analyzed (Participants) | 60 | 61
  Constipation | -0.6 (32.18) | -3.8 (34.48)
  Diarrhoea: number analyzed (Participants) | 61 | 59
  Diarrhoea | 4.4 (29.49) | 1.1 (23.95)
  Financial difficulties: number analyzed (Participants) | 61 | 60
  Financial difficulties | 0.0 (29.81) | 0.6 (24.16)

13. Secondary Outcome: Mean Change From Baseline in the EORTC Quality of Life (QOL) Questionnaire of Stomach 22 (QLQ-STO22) Scales/Items Score Scale
Description: The QLQ-STO22 consists of 22 items divided into five subscales: dysphagia, pain, reflux, eating restrictions and anxiety, as well as single items addressing dry mouth, body image, taste, and hair loss. Each item is answered on a 4-point scale, ranging from 1 (not at all) to 4 (very much). Raw scores for each subscale or single item are calculated by averaging the scores of the individual items that make up the scale. These scores are then linearly transformed to range from 0 to 100. In terms of interpretation, a higher score indicates a worse quality of life concerning the specific symptoms assessed.
Time Frame: as for outcome 12
Population: Primary Efficacy (PE) population. Only those participants contributing data at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 60 | 54
Scores on a scale
  Dysphagia scale | 3.4 (22.99) | -3.1 (16.92)
  Pain scale | -1.5 (22.20) | -0.6 (18.71)
  Reflux scale | -1.4 (21.86) | -4.1 (18.48)
  Eating restrictions scale: number analyzed (Participants) | 59 | 54
  Eating restrictions scale | 1.2 (27.83) | -3.2 (22.11)
  Anxiety scale | -2.9 (27.42) | -7.5 (24.38)
  Dry mouth scale: number analyzed (Participants) | 59 | 54
  Dry mouth scale | 2.8 (31.13) | 1.9 (32.00)
  Taste scale: number analyzed (Participants) | 59 | 51
  Taste scale | 4.5 (37.37) | 9.2 (32.03)
  Body image scale | -3.3 (37.68) | -1.9 (30.66)
  Hair loss scale: number analyzed (Participants) | 2 | 3
  Hair loss scale | -16.7 (23.57) | 0.0 (33.33)

14. Secondary Outcome: Mean Change From Baseline in Utility Score (Health Utility Index) in the EuroQoL-5 Dimensions (EQ-5D) Questionnaire
Description: The EQ-5D is a standardized instrument developed by the EuroQoL Group to measure health-related quality of life. It includes a descriptive system covering five dimensions and a Visual Analogue Scale (VAS), often referred to as the Thermometer Score.
  The Utility Score (Health Utility Index) is derived from the five dimensions of the EQ-5D descriptive system (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension has levels indicating severity (e.g., 1 = no problems, 2 = some problems, 3 = extreme problems). These combinations form a health state, which is then converted into a single index value using a country-specific value set. In the UK-based value set, the possible EQ-5D index utility values range from -0.594 to 1.0, where: 1.0 = perfect health, 0 = death and < 0 = health states considered worse than death.
Time Frame: as for outcome 12
Population: Primary Efficacy (PE) population. Only those participants contributing data at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 59 | 57
Scores on a scale | -0.17 (0.347) | -0.07 (0.328)

15. Secondary Outcome: Mean Change From Baseline in Thermometer Score (EQ VAS) in the EuroQoL-5 Dimensions (EQ-5D) Questionnaire
Description: The EQ-5D is a standardized instrument developed by the EuroQol Group to measure health-related quality of life. It includes a descriptive system covering five dimensions and a Visual Analogue Scale (VAS), often referred to as the Thermometer Score.
  The Thermometer Score is a self-rated health score using a vertical visual analogue scale , where respondents rate their overall health on a scale from 0 (worst imaginable health) to 100 (best imaginable health).
Time Frame: as for outcome 12
Population: Primary Efficacy (PE) population. Only those participants contributing data at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 61 | 60
Scores on a scale | -4.61 (23.054) | -7.90 (17.349)

16. Secondary Outcome: Percentage of Participants With Worst-case On-therapy Chemistry Toxicities
Description: The severity of chemistry parameters was graded according to NCI CTCAE version 3.0: Grade 0 (No adverse event or within normal limits), Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (life-threatening).
  Chemistry data included: Alanine aminotransferase (ALT), Albumin, Alkaline phosphatases (ALP), Aspartate aminotransferase (AST), Calcium (hypercalcemia), Calcium (hypocalcemia), Creatine Kinase (CK), Creatine, Glucose (hyperglycemia), Glucose (hypoglycemia), Magnesium (hypermagnesemia), Magnesium (hypomagnesemia), Potassium (hyperkalemia), Potassium (hypokalemia), Sodium (hypernatremia), Sodium (hyponatremia) and Total Bilirubin.
Time Frame: as for outcome 9
Population: Safety Population. Only those participants contributing data at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 260 | 262
Participants
  Alanine aminotransferase (ALT): Grade 0 | 163 | 153
  Alanine aminotransferase (ALT): Grade 1 | 87 | 94
  Alanine aminotransferase (ALT): Grade 2 | 8 | 11
  Alanine aminotransferase (ALT): Grade 3 | 2 | 4
  Alanine aminotransferase (ALT): Grade 4 | 0 | 0
  Albumin: number analyzed (Participants) | 257 | 258
  Albumin: Grade 0 | 123 | 140
  Albumin: Grade 1 | 72 | 66
  Albumin: Grade 2 | 59 | 48
  Albumin: Grade 3 | 3 | 4
  Albumin: Grade 4 | 0 | 0
  Alkaline phosphatases (ALP): number analyzed (Participants) | 260 | 260
  Alkaline phosphatases (ALP): Grade 0 | 120 | 114
  Alkaline phosphatases (ALP): Grade 1 | 113 | 109
  Alkaline phosphatases (ALP): Grade 2 | 22 | 25
  Alkaline phosphatases (ALP): Grade 3 | 5 | 12
  Alkaline phosphatases (ALP): Grade 4 | 0 | 0
  Aspartate aminotransferase (AST): Grade 0 | 108 | 93
  Aspartate aminotransferase (AST): Grade 1 | 133 | 142
  Aspartate aminotransferase (AST): Grade 2 | 16 | 21
  Aspartate aminotransferase (AST): Grade 3 | 3 | 6
  Aspartate aminotransferase (AST): Grade 4 | 0 | 0
  Calcium (hypercalcemia): number analyzed (Participants) | 256 | 262
  Calcium (hypercalcemia): Grade 0 | 237 | 242
  Calcium (hypercalcemia): Grade 1 | 17 | 19
  Calcium (hypercalcemia): Grade 2 | 2 | 1
  Calcium (hypercalcemia): Grade 3 | 0 | 0
  Calcium (hypercalcemia): Grade 4 | 0 | 0
  Calcium (hypocalcemia): number analyzed (Participants) | 256 | 262
  Calcium (hypocalcemia): Grade 0 | 129 | 134
  Calcium (hypocalcemia): Grade 1 | 74 | 81
  Calcium (hypocalcemia): Grade 2 | 50 | 43
  Calcium (hypocalcemia): Grade 3 | 3 | 4
  Calcium (hypocalcemia): Grade 4 | 0 | 0
  Creatine Kinase (CK): number analyzed (Participants) | 1 | 3
  Creatine Kinase (CK): Grade 0 | 1 | 3
  Creatine Kinase (CK): Grade 1 | 0 | 0
  Creatine Kinase (CK): Grade 2 | 0 | 0
  Creatine Kinase (CK): Grade 3 | 0 | 0
  Creatine Kinase (CK): Grade 4 | 0 | 0
  Creatinine: Grade 0 | 230 | 228
  Creatinine: Grade 1 | 21 | 33
  Creatinine: Grade 2 | 7 | 0
  Creatinine: Grade 3 | 2 | 1
  Creatinine: Grade 4 | 0 | 0
  Glucose (hyperglycemia): number analyzed (Participants) | 259 | 262
  Glucose (hyperglycemia): Grade 0 | 107 | 119
  Glucose (hyperglycemia): Grade 1 | 115 | 103
  Glucose (hyperglycemia): Grade 2 | 30 | 32
  Glucose (hyperglycemia): Grade 3 | 6 | 8
  Glucose (hyperglycemia): Grade 4 | 1 | 0
  Glucose (hypoglycemia): number analyzed (Participants) | 259 | 262
  Glucose (hypoglycemia): Grade 0 | 223 | 237
  Glucose (hypoglycemia): Grade 1 | 32 | 20
  Glucose (hypoglycemia): Grade 2 | 3 | 2
  Glucose (hypoglycemia): Grade 3 | 1 | 1
  Glucose (hypoglycemia): Grade 4 | 0 | 2
  Magnesium (hypermagnesemia): number analyzed (Participants) | 254 | 256
  Magnesium (hypermagnesemia): Grade 0 | 229 | 234
  Magnesium (hypermagnesemia): Grade 1 | 20 | 17
  Magnesium (hypermagnesemia): Grade 2 | 0 | 0
  Magnesium (hypermagnesemia): Grade 3 | 5 | 5
  Magnesium (hypermagnesemia): Grade 4 | 0 | 0
  Magnesium (hypomagnesemia): number analyzed (Participants) | 254 | 256
  Magnesium (hypomagnesemia): Grade 0 | 189 | 199
  Magnesium (hypomagnesemia): Grade 1 | 59 | 52
  Magnesium (hypomagnesemia): Grade 2 | 5 | 5
  Magnesium (hypomagnesemia): Grade 3 | 1 | 0
  Magnesium (hypomagnesemia): Grade 4 | 0 | 0
  Potassium (hyperkalemia): number analyzed (Participants) | 259 | 261
  Potassium (hyperkalemia): Grade 0 | 228 | 234
  Potassium (hyperkalemia): Grade 1 | 20 | 14
  Potassium (hyperkalemia): Grade 2 | 8 | 11
  Potassium (hyperkalemia): Grade 3 | 2 | 2
  Potassium (hyperkalemia): Grade 4 | 1 | 0
  Potassium (hypokalemia): number analyzed (Participants) | 259 | 261
  Potassium (hypokalemia): Grade 0 | 160 | 195
  Potassium (hypokalemia): Grade 1 | 75 | 54
  Potassium (hypokalemia): Grade 2 | 0 | 0
  Potassium (hypokalemia): Grade 3 | 21 | 11
  Potassium (hypokalemia): Grade 4 | 3 | 1
  Sodium (hypernatremia): number analyzed (Participants) | 259 | 261
  Sodium (hypernatremia): Grade 0 | 234 | 234
  Sodium (hypernatremia): Grade 1 | 18 | 20
  Sodium (hypernatremia): Grade 2 | 2 | 5
  Sodium (hypernatremia): Grade 3 | 3 | 2
  Sodium (hypernatremia): Grade 4 | 2 | 0
  Sodium (hyponatremia): number analyzed (Participants) | 259 | 261
  Sodium (hyponatremia): Grade 0 | 186 | 199
  Sodium (hyponatremia): Grade 1 | 52 | 42
  Sodium (hyponatremia): Grade 2 | 0 | 0
  Sodium (hyponatremia): Grade 3 | 19 | 16
  Sodium (hyponatremia): Grade 4 | 2 | 4
  Total Bilirubin: number analyzed (Participants) | 260 | 261
  Total Bilirubin: Grade 0 | 153 | 178
  Total Bilirubin: Grade 1 | 55 | 42
  Total Bilirubin: Grade 2 | 43 | 33
  Total Bilirubin: Grade 3 | 7 | 3
  Total Bilirubin: Grade 4 | 2 | 5

17. Secondary Outcome: Percentage of Participants With Worst-case On-therapy Hematologic Toxicities
Description: The severity of hematologic parameters was graded according to NCI CTCAE version 3.0: Grade 0 (No adverse event or within normal limits), Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (life-threatening).
  Hematology data included: Hemoglobin, Platelet count, Total Neutrophils (Total ANC - Total Absolute Neutrophil Count) and White Blood Cell count.
Time Frame: as for outcome 9
Population: Safety Population. Only those participants contributing data at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo
Number analyzed (Participants) | 261 | 263
Participants
  Hemoglobin: Grade 0 | 18 | 22
  Hemoglobin: Grade 1 | 104 | 121
  Hemoglobin: Grade 2 | 104 | 93
  Hemoglobin: Grade 3 | 35 | 27
  Hemoglobin: Grade 4 | 0 | 0
  Platelet count: number analyzed (Participants) | 261 | 261
  Platelet count: Grade 0 | 97 | 116
  Platelet count: Grade 1 | 95 | 86
  Platelet count: Grade 2 | 43 | 27
  Platelet count: Grade 3 | 21 | 30
  Platelet count: Grade 4 | 5 | 2
  Total Neutrophils (Total ANC - Total Absolute Neutrophil Count): number analyzed (Participants) | 240 | 249
  Total Neutrophils (Total ANC - Total Absolute Neutrophil Count): Grade 0 | 112 | 127
  Total Neutrophils (Total ANC - Total Absolute Neutrophil Count): Grade 1 | 42 | 45
  Total Neutrophils (Total ANC - Total Absolute Neutrophil Count): Grade 2 | 58 | 48
  Total Neutrophils (Total ANC - Total Absolute Neutrophil Count): Grade 3 | 22 | 27
  Total Neutrophils (Total ANC - Total Absolute Neutrophil Count): Grade 4 | 6 | 2
  White Blood Cell count: number analyzed (Participants) | 261 | 262
  White Blood Cell count: Grade 0 | 126 | 136
  White Blood Cell count: Grade 1 | 71 | 74
  White Blood Cell count: Grade 2 | 50 | 47
  White Blood Cell count: Grade 3 | 12 | 4
  White Blood Cell count: Grade 4 | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were documented from the first administration of the study medication through the end of the Long-Term Follow-up (LTFU) period, covering a duration of up to approximately 16 years. Deaths were recorded from the study initiation through the end of the LTFU period, also assessed up to approximately 16 years. On-treatment period (up to 30 days after last dose) and post-treatment follow-up phase (thereafter) are reported separately.
Description: Deaths in the Long Term Follow-up (LTFU) period were not considered adverse events. The total number at risk in the LTFU included patients who entered this period. All-cause Mortality was assessed for all participants enrolled in the study, while Serious and Other Adverse Events were assessed for all participants who received at least one dose of the study medication.
Groups:
- CapeOx Plus Lapatinib: CapeOx plus Lapatinib combination therapy: Events up to 30 days post-treatment
- CapeOx Plus Placebo: CapeOx plus Placebo combination therapy: Events up to 30 days post-treatment
- CapeOx Plus Lapatinib (Long Term Follow-up (LTFU)): CapeOx plus Lapatinib combination therapy (Long Term Follow-up (LTFU)): Deaths in the Long Term Follow-up (LTFU) period were not considered adverse events.
- CapeOx Plus Placebo (Long Term Follow-up (LTFU)): CapeOx plus Placebo combination therapy (Long Term Follow-up (LTFU)): Deaths in the Long Term Follow-up (LTFU) period were not considered adverse events.
Arm/Group | CapeOx Plus Lapatinib | CapeOx Plus Placebo | CapeOx Plus Lapatinib (Long Term Follow-up (LTFU)) | CapeOx Plus Placebo (Long Term Follow-up (LTFU))
All-Cause Mortality (participants affected / at risk) | 42/272 | 40/273 | 199/230 | 189/233
Serious Adverse Events (participants affected / at risk) | 73/270 | 54/267 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 243/270 | 214/267 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CapeOx Plus Lapatinib (N=270) | CapeOx Plus Placebo (N=267) | CapeOx Plus Lapatinib (Long Term Follow-up (LTFU)) (N=0) | CapeOx Plus Placebo (Long Term Follow-up (LTFU)) (N=0)
Anaemia (Blood and lymphatic system disorders) | 7 | 4 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | NA | NA
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | NA | NA
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | NA | NA
Atrial fibrillation (Cardiac disorders) | 2 | 0 | NA | NA
Cardiac tamponade (Cardiac disorders) | 1 | 0 | NA | NA
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | NA | NA
Left ventricular dysfunction (Cardiac disorders) | 2 | 0 | NA | NA
Pericardial effusion (Cardiac disorders) | 0 | 1 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 1 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 16 | 1 | NA | NA
Dysphagia (Gastrointestinal disorders) | 2 | 1 | NA | NA
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0 | NA | NA
Gastric dilatation (Gastrointestinal disorders) | 0 | 1 | NA | NA
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 2 | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2 | NA | NA
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | NA | NA
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | NA | NA
Haematemesis (Gastrointestinal disorders) | 0 | 2 | NA | NA
Ileus spastic (Gastrointestinal disorders) | 0 | 1 | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1 | NA | NA
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | NA | NA
Melaena (Gastrointestinal disorders) | 1 | 1 | NA | NA
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Nausea (Gastrointestinal disorders) | 6 | 2 | NA | NA
Obstruction gastric (Gastrointestinal disorders) | 1 | 1 | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | NA | NA
Vomiting (Gastrointestinal disorders) | 7 | 6 | NA | NA
Asthenia (General disorders) | 2 | 4 | NA | NA
Condition aggravated (General disorders) | 0 | 1 | NA | NA
Death (General disorders) | 2 | 0 | NA | NA
Drowning (General disorders) | 0 | 1 | NA | NA
Fatigue (General disorders) | 3 | 0 | NA | NA
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | NA | NA
Oedema peripheral (General disorders) | 1 | 0 | NA | NA
Pyrexia (General disorders) | 4 | 1 | NA | NA
Sudden death (General disorders) | 1 | 0 | NA | NA
Jaundice (Hepatobiliary disorders) | 1 | 0 | NA | NA
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | NA | NA
Contrast media reaction (Immune system disorders) | 1 | 0 | NA | NA
Drug hypersensitivity (Immune system disorders) | 1 | 0 | NA | NA
Abdominal infection (Infections and infestations) | 1 | 0 | NA | NA
Bacteraemia (Infections and infestations) | 1 | 0 | NA | NA
Cellulitis (Infections and infestations) | 0 | 1 | NA | NA
Gastroenteritis (Infections and infestations) | 1 | 0 | NA | NA
Gastrointestinal infection (Infections and infestations) | 0 | 1 | NA | NA
Herpes zoster (Infections and infestations) | 0 | 1 | NA | NA
Large intestine infection (Infections and infestations) | 0 | 1 | NA | NA
Lung abscess (Infections and infestations) | 0 | 1 | NA | NA
Peritonitis (Infections and infestations) | 0 | 1 | NA | NA
Pneumonia (Infections and infestations) | 6 | 3 | NA | NA
Pneumonia aspiration (Infections and infestations) | 2 | 0 | NA | NA
Sepsis (Infections and infestations) | 1 | 1 | NA | NA
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | NA | NA
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Spinal cord injury thoracic (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Alanine aminotransferase increased (Investigations) | 0 | 1 | NA | NA
Blood bilirubin increased (Investigations) | 0 | 1 | NA | NA
Ejection fraction decreased (Investigations) | 1 | 1 | NA | NA
Haemoglobin decreased (Investigations) | 1 | 0 | NA | NA
Liver function test abnormal (Investigations) | 0 | 1 | NA | NA
Platelet count decreased (Investigations) | 1 | 0 | NA | NA
Weight decreased (Investigations) | 0 | 1 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | NA | NA
Dehydration (Metabolism and nutrition disorders) | 6 | 1 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Aphasia (Nervous system disorders) | 1 | 0 | NA | NA
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | NA | NA
Dizziness (Nervous system disorders) | 1 | 0 | NA | NA
Epilepsy (Nervous system disorders) | 1 | 0 | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | NA | NA
Nervous system disorder (Nervous system disorders) | 1 | 0 | NA | NA
Paraesthesia (Nervous system disorders) | 1 | 0 | NA | NA
Seizure (Nervous system disorders) | 0 | 1 | NA | NA
Speech disorder (Nervous system disorders) | 1 | 0 | NA | NA
Syncope (Nervous system disorders) | 0 | 1 | NA | NA
Device occlusion (Product Issues) | 0 | 1 | NA | NA
Confusional state (Psychiatric disorders) | 0 | 1 | NA | NA
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | NA | NA
Oliguria (Renal and urinary disorders) | 1 | 0 | NA | NA
Renal failure (Renal and urinary disorders) | 1 | 0 | NA | NA
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | NA | NA
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Circulatory collapse (Vascular disorders) | 1 | 0 | NA | NA
Deep vein thrombosis (Vascular disorders) | 1 | 0 | NA | NA
Haemorrhage (Vascular disorders) | 1 | 0 | NA | NA
Venous thrombosis (Vascular disorders) | 1 | 0 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CapeOx Plus Lapatinib (N=270) | CapeOx Plus Placebo (N=267) | CapeOx Plus Lapatinib (Long Term Follow-up (LTFU)) (N=0) | CapeOx Plus Placebo (Long Term Follow-up (LTFU)) (N=0)
Abdominal distension (Gastrointestinal disorders) | 16 | 9 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 27 | 32 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 20 | 27 | NA | NA
Constipation (Gastrointestinal disorders) | 30 | 54 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 146 | 77 | NA | NA
Dyspepsia (Gastrointestinal disorders) | 14 | 20 | NA | NA
Nausea (Gastrointestinal disorders) | 128 | 113 | NA | NA
Stomatitis (Gastrointestinal disorders) | 19 | 10 | NA | NA
Vomiting (Gastrointestinal disorders) | 116 | 93 | NA | NA
Asthenia (General disorders) | 46 | 36 | NA | NA
Fatigue (General disorders) | 64 | 60 | NA | NA
Oedema peripheral (General disorders) | 14 | 18 | NA | NA
Pyrexia (General disorders) | 30 | 26 | NA | NA
Weight decreased (Investigations) | 43 | 33 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 107 | 85 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 16 | NA | NA
Dizziness (Nervous system disorders) | 14 | 14 | NA | NA
Headache (Nervous system disorders) | 7 | 14 | NA | NA
Neuropathy peripheral (Nervous system disorders) | 53 | 58 | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 34 | 29 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 19 | NA | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 57 | 40 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 5 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 46 | 16 | NA | NA
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 16 | 7 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.